CLINICAL TRIAL: NCT01262404
Title: Imaging Cerebral and Sub-cerebral Correlates of Meditative States
Acronym: calm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston University (Other)
Collaborators: Emory University (Other)
Responsible Party: Professor Eric L. Schwartz, Boston University
Other Study IDs: BU-Emory-01; AT005728-01 (Other Grant/Funding Number: NCCAM)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HealthEd,Minfdulness,Compassion: HealthEd receives training health education. Mindfulness receives training in mindfulness meditation. Compassion receives training in compassion meditation.

SUMMARY:
Three groups of subjects are trained to practice mindfulness meditation, compassion meditation, or attend a health training control class. Individuals from each group will undergo structural and functional brain imaging before and after training. The hypothesis is that the compassion meditation group will show the largest changes in brain structure and function. In a second series of experiments, the subjects practicing a Tibetan meditation practice will be undergo MRI thermometry imaging to construct detailed three dimensional temperature maps of their bodies before, during, and after they perform this practice.

DETAILED DESCRIPTION:
Structural (MRI) Imaging will be used to measure changes in cortical thickness in the pre and post training groups. Function (fMRI) Imaging will be used to measure changes in cortical and sub-cortical responses to a series of affectively controlled visual images, presented during scanning. MRI Thermometry Imaging will be used to construct three dimensional temperature maps of subjects while performing meditation in the scanner.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 for the mindfulness-compassion study
* Prior training in gtummo meditation for the gtummo study

Exclusion Criteria:

* Previous experience with meditation for the mindfulness-compassion study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Schwartz, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Dept. of Cognitive and Neural Systems, Boston, Massachusetts, United States